CLINICAL TRIAL: NCT01622283
Title: Pharmacokinetic Study of Levocetirizine Oral Solution-An Open-label, Randomized, Cross-over Study to Evaluate the Pharmacokinetics, the Safety and Tolerability of Levocetirizine Oral Solution (5 mg) and Cetirizine Dry Syrup (10 mg), Following a Single Dose in Japanese Healthy Male Subjects-
Brief Title: Pharmacokinetic Study of Levocetirizine Oral Solution
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 116459
Record Dates: First submitted 2012-04-19; First posted 2012-06-19 (Estimated); Last update posted 2017-06-12 (Actual); Status verified 2017-06

CONDITIONS: Rhinitis, Allergic, Perennial and Seasonal
MeSH Terms: conditions — Rhinitis | interventions — levocetirizine; Cetirizine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Levocetirizine oral solution 5 mg (Experimental): Levocetirizine oral solution 5 mg
  Interventions: Drug: Levocetirizine
- Cetirizine dry syrup 10 mg (Active Comparator): Cetirizine dry syrup 10 mg
  Interventions: Drug: Cetirizine

INTERVENTIONS:
Drug: Levocetirizine — Levocetirizine
  Arms: Levocetirizine oral solution 5 mg
Drug: Cetirizine — Cetirizine
  Arms: Cetirizine dry syrup 10 mg

SUMMARY:
This study will be a single center, open-label, randomized, single dose, in the fasted condition and 2-way crossover study to evaluate the pharmacokinetics, the safety and tolerability of levocetirizine oral solution 5 mg and cetirizine dry syrup 10 mg in Japanese healthy male subjects.

Approximately 20 subjects will receive both treatments of levocetirizine oral solution 5 mg and cetirizine dry syrup 10 mg in the design. Serial pharmacokinetic samples will be collected and safety assessments will be performed following each dose.

The primary objective of the study is to demonstrate the bioequivalence of levocetirizine in plasma, when given as levocetirizine oral solution 5 mg relative to cetirizine DS 10 mg in Japanese healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring. A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the Investigator and the GSK Medical Monitor agree that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Japanese male between 20 and 55 years of age inclusive, at the time of signing the informed consent.
* Non-smoker or ex-smoker having ceased smoking for at least 6 months.
* Body weight => 50 kg and BMI within the range 18.5 - 25.0 kg/m2 at screening.
* A signed and dated written informed consent is obtained from the subject.
* Able to complete all study procedures and planned treatment periods.
* ALT, alkaline phosphatase and bilirubin =< 1.5xULN (isolated bilirubin > 1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin < 35%).
* Single QTcB < 450 msec at screening.

Exclusion Criteria:

* The subject is positive for syphilis, Hepatitis B surface antigen, Hepatitis C antibody, HIV1/2 antibody, or HTLV-1 antibody at screening.
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* The subject has a history of allergic rhinitis.
* The subject is currently participating in another clinical study or post-marketing study in which the subject is or will be exposed to an investigational or a non-investigational drug or device.
* The subject has a history or current conditions of drug abuse or alcoholism.
* A positive pre-study drug screen.
* History of regular alcohol consumption within 6 months of the study defined as an average weekly intake of >14 drinks. One drink is equivalent to 12 g of alcohol: 12 ounces (350 mL) of beer, 5 ounces (150 mL) of wine or 1.5 ounces (45 mL) of 80 proof distilled spirits.
* The subject has participated in a clinical trial and has received an investigational product or a non-investigational drug within 4 months prior to the first dosing day in the current study.
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Unable to refrain from the use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 14 days or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy.
* Where participation in the study would result in donation of blood or blood products => 400 mL within 3 months or => 200 mL within 1 month.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* Subject is mentally or legally incapacitated.

Ages: 20 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2012-05-02 (Actual); Primary Completion 2012-06-10 (Actual); Study Completion 2012-06-10 (Actual)

PRIMARY OUTCOMES:
AUC(0-48) of levocetirizine | pre, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12, 16, 24, 36, 48h post dose
  AUC(0-48): Area under plasma concentration time curve from pre-dose to 48h.
Cmax of levocetirizine | pre, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12, 16, 24, 36, 48h post dose
  Cmax: Maximum observed concentration.

SECONDARY OUTCOMES:
Adverse events | up to 48h post dose
  Number of participants with adverse events as a measure of safety and tolerability.
Safety and tolerability | up to 48h post dose
  Safety and tolerability of levocetirizine and cetirizine in terms of clinical laboratory tests, vital sign, body weight and ECG.
Vital sign | up to 48h post dose
  Systolic and diastolic blood pressure, body temperature and pulse rate.
Body weight | up to 48h post dose
ECG | up to 48h post dose
  Heart rate, PR, QRS, QT, and QTc intervals.
Laboratory tests | up to 48h post dose
  Clinical Chemistry (Total Protein, Albumin, Total and Direct Bilirubin, BUN, Creatinine, Uric Acid, TG, Total Cholesterol, LDL and HDL-cholesterol, AST, ALT, Alkaline Phosphatase, LDH, GGT, CPK, Amylase, Glucose(fasting), Sodium, Potassium, Chloride, Calcium, Phosphorus), Hematology (Platelet Count, RBC Count, WBC Count (absolute), Reticulocyte Count, Hemoglobin, Hematocrit, RBC Indices (MCV, MCH, MCHC) and Automated WBC Differential (Neutrophils, Lymphocytes, Monocytes, Eosinophils, Basophils)) and Urinalysis (Specific Gravity, pH, Glucose, Protein, Blood, Ketones and Microscopic Examination)
AUC(0-inf), MRT, tmax, and t1/2 of levocetirizine | pre, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12, 16, 24, 36, 48h post dose
  AUC(0-inf): Area under the concentration-time curve from time pre-dose extrapolated to infinite time, MRT: Mean residence time, tmax: Time of occurrence of Cmax, and t1/2: Terminal phase half-life.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Kagoshima, Japan

REFERENCES:
- [Derived] Ino H, Hara K, Honma G, Doi Y, Fukase H. Comparison of levocetirizine pharmacokinetics after single doses of levocetirizine oral solution and cetirizine dry syrup in healthy Japanese male subjects. J Drug Assess. 2014 Jun 3;3(1):38-42. doi: 10.3109/21556660.2014.928302. eCollection 2014. PMID 27536452
- See also: Results for study 116459 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/116459?search=study&study_ids=116459#rs